CLINICAL TRIAL: NCT03182920
Title: Effect of Age on the Pharmacokinetics, Safety, and Tolerability of Lasmiditan in Healthy Subjects
Brief Title: A Study of Lasmiditan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16852; H8H-MC-LAHA (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2019-12-06 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Intervention Model Description: 2 Groups: Group 1 - Double-blind Randomized 2-Period Crossover, Group 2 - Open-label single dose
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 200 mg Lasmiditan (Group 1 Elderly) (Experimental): 200 milligrams (mg) lasmiditan on Day 1 of 1 of 2 dosing periods.
  Interventions: Drug: Lasmiditan
- Placebo (Group 1 Elderly) (Placebo Comparator): Placebo on Day 1 of 1 of 2 dosing periods.
  Interventions: Drug: Placebo
- 200 mg Lasmiditan (Group 2 Young) (Experimental): 200 mg lasmiditan on Day 1.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Oral administration
  Other Names: LY573144
  Arms: 200 mg Lasmiditan (Group 1 Elderly); 200 mg Lasmiditan (Group 2 Young)
Drug: Placebo — Oral administration
  Arms: Placebo (Group 1 Elderly)

SUMMARY:
The purpose of this study is to look at the amount of study drug that gets into the blood stream and how long it takes the body to get rid of it by comparing the results of healthy elderly participants to those of healthy young participants. The tolerability of the study drug will be evaluated. Information about any side effects that may occur will also be collected.

This study will last up to approximately 19 days, not including screening. This study requires either one (Group 2) or two (Group 1) stays at the clinic each of at least four days/three nights. Participants will return for a follow-up seven days after last dose of study drug. Screening is required within 28 days prior to Day 1.

This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination.
* Have a body mass index (BMI) of 19 to 35 kilograms per meter squared (kg/m²) inclusive, at the time of screening.

Exclusion Criteria:

* Have known allergies to lasmiditan, related compounds or any components of the formulation.
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study.
* Show evidence of active renal disease or estimated glomerular filtration rate (eGFR) less than 60 milliliter per minute (mL/min) per 1.73 m².
* Show evidence of or positive serology for human immunodeficiency virus (HIV) infection, hepatitis B or C.
* Are women with a positive pregnancy test or women who are lactating.
* Have a clinically significant abnormality in the neurological examination.
* Have a history of syncope, presyncopy, uncontrolled vertigo, postural dizziness, or at risk for falls, as judged to be clinically significant by the investigator.
* Have orthostatic hypotension with or without dizziness and/or syncope at screening or Day -1 upon repeat testing, or a history of it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Daytona Beach, Daytona Beach, Florida
  - Covance Evansville, Evansville, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Group 1 Elderly: Placebo on day 1 of period 1 200 mg of lasmiditan on Day 1 of period 2.
- Sequence 2: Group 1 Elderly: 200 mg of lasmiditan on Day 1 of period 1. Placebo on Day 1 of period 2.
- 200 mg Lasmiditan (Group 2 Young): 200 mg of lasmiditan on Day 1.
Period: Period 1
Arm/Group | Sequence 1: Group 1 Elderly | Sequence 2: Group 1 Elderly | 200 mg Lasmiditan (Group 2 Young)
Started | 9 | 9 | 17
Completed | 9 | 9 | 17
Not Completed | 0 | 0 | 0
Period: Washout Period
Arm/Group | Sequence 1: Group 1 Elderly | Sequence 2: Group 1 Elderly | 200 mg Lasmiditan (Group 2 Young)
Started | 9 | 9 | 0
Completed | 9 | 9 | 0
Not Completed | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: Group 1 Elderly | Sequence 2: Group 1 Elderly | 200 mg Lasmiditan (Group 2 Young)
Started | 9 | 9 | 0 (Young participants on Lasmiditan did not move to study period 2.)
Completed | 9 | 9 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Group 1 Elderly: Placebo on Day 1 of 1 of 2 dosing periods or 200 milligrams (mg) lasmiditan on Day 1 of 1 of 2 dosing periods.
- Total: Total of all reporting groups
Arm/Group | Group 1 Elderly | 200 mg Lasmiditan (Group 2 Young) | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (5.4) | 31.3 (7.7) | 51.5 (21.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 18 | 12 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 17 | 34
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Lasmiditan
Description: Maximum Observed Drug Concentration (Cmax) of Lasmiditan.
Time Frame: Day 1:Predose,0.5, 1, 1.5,2, 2.5, 3, 4,6, 8, 12 hours; Day 2: 24,36 hours; Day 3:48 hours
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms Per Millilitre (ng/mL)
Groups:
- 200 mg Lasmiditan (Group 1 Elderly): 200 mg lasmiditan on Day 1 of 1 of 2 dosing periods.
Arm/Group | 200 mg Lasmiditan (Group 1 Elderly) | 200 mg Lasmiditan (Group 2 Young)
Number analyzed (Participants) | 18 | 17
Nanograms Per Millilitre (ng/mL) | 368 (43) | 304 (40)
Statistical Analysis 1: Comparison: 200 mg Lasmiditan (Group 1 Elderly) vs 200 mg Lasmiditan (Group 2 Young); Test type: Superiority; Ratio of geometric least squares means = 1.21, 90% CI 2-sided [0.962 to 1.52]

2. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Lasmiditan
Description: Area under the concentration versus time curve from zero to infinity
Time Frame: Day 1:Predose,0.5, 1, 1.5,2, 2.5, 3, 4,6, 8, 12 hours; Day 2: 24,36 hours; Day 3:48 hours
Population: All participants who received at least one dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms*hour per Millilitre (ng.h/mL)
Arm/Group | 200 mg Lasmiditan (Group 1 Elderly) | 200 mg Lasmiditan (Group 2 Young)
Number analyzed (Participants) | 18 | 17
Nanograms*hour per Millilitre (ng.h/mL) | 2480 (44) | 1970 (30)
Statistical Analysis 1: Comparison: 200 mg Lasmiditan (Group 1 Elderly) vs 200 mg Lasmiditan (Group 2 Young); Test type: Superiority; Ratio of geometric least squares means = 1.26, 90% CI 2-sided [1.03 to 1.55]

ADVERSE EVENTS:
Time Frame: Up to 10 Days
Arm/Group | Placebo (Group 1 Elderly) | 200 mg Lasmiditan (Group 1 Elderly) | 200 mg Lasmiditan (Group 2 Young)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 3/18 | 8/18 | 8/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Group 1 Elderly) (N=18) | 200 mg Lasmiditan (Group 1 Elderly) (N=18) | 200 mg Lasmiditan (Group 2 Young) (N=17)
Photopsia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sensation of foreign body (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03182920/SAP_000.pdf
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT03182920/Prot_002.pdf